CLINICAL TRIAL: NCT07369063
Title: Impact of Vitamin D Therapy on Thyroid Function and Antibody Levels in Pediatric Graves' Disease: A Pilot Feasibility Trial
Brief Title: Impact of Vitamin D Therapy on Thyroid Function and Antibody Levels in Pediatric Graves' Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 25-0285
Record Dates: First submitted 2025-07-14; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Graves Disease; Graves' Disease; Hyperthyroidism
Keywords: vitamin d; graves disease; hyperthyroidism
MeSH Terms: conditions — Graves Disease; Hyperthyroidism | interventions — Ergocalciferols; Methimazole

STUDY DESIGN:
Intervention Model Description: The control group receives standard methimazole therapy and has the option of taking up to 1000 IU/day of over-the-counter vitamin D2, which is not provided by the study. This is to ensure ethical considerations related to vitamin D deficiency are met while maintaining a comparison group. Should the patients in the control group have vitamin D levels <20 ng/mL, patients will be strongly advised to take the 1000 IU of vitamin D daily for repletion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- High-Dose Vitamin D2 + Methimazole (Experimental): Participants in this arm will receive methimazole at a dose determined by their treating physician, according to standard clinical practice guidelines for pediatric Graves' disease. In addition, they will receive high-dose vitamin D2 (ergocalciferol) 50,000 IU orally weekly for the first 8 weeks, followed by 50,000 IU orally every two weeks for the remaining 16 weeks of the study.
  Interventions: Drug: Ergocalciferol 50,000 IU; Drug: Methimazole
- Methimazole (with optional low dose Vitamin D2) (Placebo Comparator): Participants in this arm will receive methimazole at a dose determined by their treating physician, according to standard clinical practice guidelines for pediatric Graves' disease. Participants will have the option of taking up to 1000 IU of vitamin D2 daily, purchased over-the-counter, but this will not be provided by the study. This is to address potential vitamin D deficiency while maintaining a comparison group.
  Interventions: Drug: Methimazole

INTERVENTIONS:
Drug: Ergocalciferol 50,000 IU — Participants will receive ergocalciferol 50,000 IU oral capsules weekly for the first 8 weeks, followed by 50,000 IU every two weeks for the subsequent 16 weeks (total 24 weeks).
  Arms: High-Dose Vitamin D2 + Methimazole
Drug: Methimazole — Methimazole is considered standard of care for pediatric Graves' disease. Dosing is determined and adjusted by the participant's treating physician

SUMMARY:
The goal of this randomized pilot feasibility clinical trial is to determine the feasibility of implementing a protocol for a larger trial to assess the effects of high-dose vitamin D supplementation in pediatric patients (9-17 years old) newly diagnosed with Graves' disease. The main questions it aims to answer are:

What are the recruitment and adherence rates for a larger trial using this protocol? Is the data collection process complete and robust enough for a larger trial? What are the potential barriers to implementing a larger-scale trial? Researchers will compare vitamin D supplementation plus standard methimazole therapy to methimazole therapy alone (with participants permitted to take up to 1000 International Units of vitamin D2 daily) to explore potential effects on thyroid hormone and antibody levels.

Participants will:

Be randomized to either the intervention or control group. Take study medications (vitamin D or placebo) as directed. Attend regular study visits for blood tests and clinical assessments. Complete medication logs.

DETAILED DESCRIPTION:
This pilot feasibility study will evaluate the practicality of conducting a larger randomized controlled trial (RCT) investigating the impact of high-dose vitamin D2 (ergocalciferol) supplementation as an adjunctive therapy to standard methimazole treatment in pediatric patients aged 9-17 years newly diagnosed with Graves' disease (GD). This study aims to address the current gap in research regarding vitamin D supplementation's effect on antibody and thyroid hormone trends in this population. Specifically, the study will examine the feasibility of recruitment, adherence to the intervention regimen, completeness of data collection, and any potential barriers to implementing a larger-scale trial.

The rationale for this study stems from the observed association between low vitamin D levels and an increased risk of Graves' disease, coupled with the limited data on vitamin D supplementation's influence on disease progression in children. This pilot study will investigate whether high-dose vitamin D supplementation, alongside methimazole, affects Thyroid Receptor Antibody (TRAb) and Thyroid Stimulating Immunoglobulin (TSI) antibody levels, as well as thyroid hormone levels (Total T3, Free Thyroxine, Total Thyroxine, TSH), in newly diagnosed pediatric GD patients.

Participants will be randomized 1:1 to either an intervention arm (methimazole + high-dose vitamin D2) or a control arm (methimazole only, with the option of taking up to 1000 IU/day of vitamin D2). The intervention arm will receive 50,000 IU of vitamin D2 weekly for 8 weeks, followed by 50,000 IU every two weeks for 16 weeks, along with standard methimazole therapy as directed by their treating endocrinologist. The control arm will receive standard methimazole therapy alone, per their physician's orders, with the option of taking up to 1000 IU of Over-the-counter (OTC) vitamin D2 daily, if desired. The study will not provide this OTC vitamin D.

The primary feasibility outcomes will be: (1) recruitment rate; (2) adherence rate to the vitamin D supplementation, assessed through pill counts, medication logs, and self-report; (3) data completeness; and (4) identification of any barriers encountered during study implementation. Exploratory clinical outcomes will include time to normalization of thyroid function tests and the percentage change from baseline in TRAb and TSI antibody levels at 24 weeks. Safety and tolerability will be closely monitored, with particular attention to hypercalcemia and hypervitaminosis D. Data on adverse events will be collected and graded using the CTCAE v5.0.

Data analysis will primarily focus on descriptive statistics for feasibility outcomes. Exploratory clinical outcomes will be analyzed to estimate effect sizes and variability, informing the design of a future, adequately powered RCT. This pilot study is not powered to detect statistically significant differences in clinical outcomes.

This study will provide critical preliminary data and feasibility metrics to inform the development of a larger, more definitive RCT evaluating vitamin D's efficacy as an adjunctive therapy in pediatric Graves' disease. This research has the potential to significantly advance our understanding of the role of vitamin D in autoimmune thyroid disease and contribute to improved treatment strategies for children with Graves' disease.

The FDA has granted an Investigational New Drug (IND) exemption (PIND 176865, dated April 30, 2025) for this pilot feasibility study evaluating high-dose vitamin D2 in children with Graves' disease. The exemption allows the study to proceed without a full IND application.

ELIGIBILITY:
Inclusion Criteria:

* All new pediatric participants aged 9-17 years with a new diagnosis of GD who will be started on methimazole, will be offered to participate at the time of diagnosis.
* Biochemical features include:
* Suppressed TSH <0.1.
* Elevated T3
* Elevated Free T4
* Elevated T4
* Positive TSI or TRAb. The presence of antibodies is diagnostic.
* Our study will offer enrollment to non-English speaking participants

Exclusion Criteria:

* Initial hydroxy vitamin D levels >80 ng/mL
* Hypocalcemia, corrected calcium based on albumin <8.4 mg/dL
* Hypercalcemia, corrected calcium based on albumin >10.5 mg/dL
* Conditions that affect vitamin D metabolism such as: malabsorption, chronic kidney or liver disease, nephrocalcinosis, hyperparathyroidism
* Current use of medications which are known to affect thyroid function or vitamin D metabolism such as thyroid hormone replacement, corticosteroids, anticonvulsants
* Allergy to vitamin D or methimazole
* Diagnosis of Hashitoxicosis or thyrotoxicosis (both TSH receptor antibody (TRAb) and thyroid-stimulating immunoglobulin (TSI) levels are negative)
* Participants under the age of 9 years at the time of diagnosis
* Pregnant participants
* Active or uncontrolled infections, other significant medical conditions deemed by the investigator to interfere with study participation or pose undue risk to the participant.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Feasibility Metrics: Recruitment Rate | through study completion, an average of 1 yea
  Percentage of eligible participants approached who consent to participate in the study. This metric will assess the efficiency of recruitment strategies.
Feasibility Metrics: Adherence Rate | From enrollment to 24 week/6month follow up visit
  Percentage of prescribed vitamin D doses taken by participants in the intervention arm. Adherence will be tracked via pill counts and participant self-report.
Feasibility Metrics: Data Completeness | From baseline data collection to the 24-week/6-month follow-up visit.
  Percentage of completed data fields for key outcome measures (thyroid function tests, TSI levels, etc.). This will assess the quality and completeness of data collection.
Feasibility Metrics: Implementation Barriers | through study completion, an average of 1 year
  A qualitative assessment of any challenges encountered during the study implementation (e.g., recruitment difficulties, adherence issues, logistical problems). This assessment will inform strategies for overcoming these barriers in a future, larger-scale RCT.

SECONDARY OUTCOMES:
Time to Normalization and Thyroid function Trends | from enrollment to 24 week/6month follow up visit
  We hypothesize that patients receiving high-dose vitamin D will achieve normal TSH, T3, Free T4 and T4 levels significantly faster than those receiving methimazole alone. Thyroid function tests will be measured at baseline, 6, 12 and 24 weeks, and time to normalization will be compared between groups.

OTHER OUTCOMES:
Change in TRAb and TSI Levels | from enrollment to 24 week/6month visit
  We hypothesize that patients receiving high-dose vitamin D will experience a significantly greater percentage reduction in TSH R-Ab and TSI levels at 24 weeks compared to those receiving methimazole alone. Antibody levels will be measured at baseline and 24 weeks, and the percentage change from baseline will be compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Hyman, MD, Principal Investigator — Northwell Health
Locations (1):
- Pediatric Endocrinology at Northwell Health, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data from this pilot feasibility study will not be shared immediately due to the small sample size and the increased risk of participant re-identification. However, data sharing aligned with journal requirements will be considered upon publication of the study results. A detailed data sharing plan will be developed at that time, addressing ethical considerations and ensuring participant privacy while maximizing the scientific value of the data. This plan will outline the specific data to be shared (e.g., de-identified data, specific variables) and the process for requesting access.
Supporting Information: Study Protocol, SAP
Time Frame: Data sharing will be considered upon acceptance of the manuscript for publication in a peer-reviewed journal.
Access Criteria: Researchers may request access to the de-identified individual participant data by contacting Dr Sharon Hyman or Dr Sofya Ilmer. Requests will be reviewed based on scientific merit, adherence to data use agreements, and capacity to protect participant confidentiality. A data use agreement will be required. Data will be shared in a format compliant with relevant privacy regulations (e.g., HIPAA).

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan: Study protocol and Statistical Analysis (2025-06-26): https://cdn.clinicaltrials.gov/large-docs/63/NCT07369063/Prot_SAP_000.pdf
  • Study Protocol: FDA IND exemption (2025-04-30): https://cdn.clinicaltrials.gov/large-docs/63/NCT07369063/Prot_001.pdf
  • Informed Consent Form: Consent form guardian or adult (2025-06-26): https://cdn.clinicaltrials.gov/large-docs/63/NCT07369063/ICF_002.pdf
  • Informed Consent Form: assent form for child (2025-06-26): https://cdn.clinicaltrials.gov/large-docs/63/NCT07369063/ICF_003.pdf